CLINICAL TRIAL: NCT01271335
Title: Collagenase Total Occlusion-1 Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Bradley Strauss, Chief of the Schulich Heart Program, Head of the Division of Cardiology and Reichmann Chair in Cardiovascular Science, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO-1; CIHR (Other Grant/Funding Number: Canadian Institutes for Health Research)
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Total Occlusions
Keywords: CTO; Angioplasty; PCI
MeSH Terms: interventions — Collagenases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Collagenase (MZ-004) (Experimental): Local intra-coronary administration of MZ-004 at or into the CTO
  Interventions: Biological: collagenase

INTERVENTIONS:
Biological: collagenase — Lyophilized powder / sterile dosage form for single local intravascular administration via the occluded coronary.
  Other Names: MZ-004

SUMMARY:
A prospective, three-center, phase I safety and tolerability dose escalation study, evaluating 28 subjects in 4 discrete dose cohorts of acute intracoronary injected collagenase ranging from 300 - 1200 µg prior to routine standard-of-care percutaneous revascularization procedures in subjects with chronic total coronary artery occlusions (CTOs).

DETAILED DESCRIPTION:
Enrolment is expected to occur over 24 months with total study duration of approximately 30 months. Five (5) subjects will be enrolled into each dose cohort. The dose cohorts will be studied in a sequential fashion, starting with the lowest doses and escalating to the highest doses. It is anticipated that each subject's involvement with the study will be 3.5 months. In addition, eight (8) subjects will be included in the highest dose cohort to collect pharmacokinetic plasma samples.

Subject enrollment and dosing within each dose cohort will be staged such that the next subsequent subject will not be dosed until the previous subject has been successfully discharged from the hospital after the angioplasty attempt. At a minimum there will be 3 days in between each subject dosing to ensure product safety.

There will be no advancement to the higher dose cohort until all 5 subjects have been discharged from the hospital and a safety review is conducted by the Data Safety Monitoring Board (DSMB) on the cardiac safety measures and the treatment deemed safe to proceed to the next dosing level.

A total of 28 male and / or female subjects suffering from CAD with a CTO will be enrolled into the study at three sites (Sunnybrook Health Sciences Centre and St. Michael's Hospital, Toronto, Ontario, and and Laval Hospital Research Centre, Quebec City, Quebec,Canada). All subjects will have had one or more previous failed angioplasty attempt(s) of the occluded artery. Subjects who have signed an Informed Consent Form (ICF) and meeting all inclusion criteria and having none of the exclusion criteria at Visit 1 (Screening) will be included in the study. All potentially enrollable subjects at Sunnybrook will be reviewed by either of two cardiologist not involved in the study to discuss the available options for the subject and to approve enrollment decisions. Eligible subjects that agree to participate will be treated in a two part procedure. On Day0 using standard angioplasty techniques to access the specified occluded coronary artery, Collagenase (MZ-004) will be directly injected into the occluded artery through a microcatheter that has been positioned immediately adjacent to or into the proximal cap of the occlusion. The catheters and arterial sheath will then be removed and the subject will be monitored overnight on the ward. The following day (Day1), the subject will be brought back to the catheterization laboratory and undergo an angioplasty using standard angioplasty techniques. Routine post-procedural management will then be followed. The subject will be discharged on Day2 in the absence of any cardiac complications (such as elevated cardiac enzymes or large pericardial effusion as judged by the Investigator and determined by echocardiography). Prior to the angioplasty procedure on Day1 and again on Day2 prior to discharge, the subject will undergo an echocardiogram to determine the presence and severity of a pericardial effusion. A moderate or large pericardial effusion or any sign of tamponade on Day1 will be a contraindication to performing the procedure, and the subject will be terminated from the study. A telephone follow-up will be performed 30 days post Day1 in all subjects who have signed an ICF and been enrolled in the study. At 3 months, subjects will undergo an outpatient coronary Computer Tomography (CT) angiogram to ensure there are no delayed effects on the treated vessel (e.g. aneurysm formation), the myocardium or the pericardium.

The primary objective is to evaluate the safety and tolerability of acute intracoronary doses of collagenase (MZ-004) in symptomatic subjects with coronary CTO.

The secondary objective is to obtain preliminary efficacy information of guidewire crossing with increasing doses of intracoronary collagenase in subjects with previously failed at least one previous attempt in coronary CTO.

ELIGIBILITY:
Inclusion Criteria:

Candidates for this study must meet ALL of the following inclusion criteria:

* Subject is willing and able to provide an informed consent
* Subject is willing and able to comply with the study procedures and follow-up
* Subject is 35 years of age or older
* Women who are non-reproductive, or reproductive women who are willing and able to practice effective birth control methods. A urine pregnancy test should be done at the screening/Day0 on all reproductive women of child bearing ability
* Subjects with CTO (older than 6 weeks or unknown duration based on the investigator's assessment of appropriateness for the study) with a clinical indication for revascularization. In subjects with occlusions of unknown duration, there must be absence of any identifiable ischemic event in the 6 weeks prior to enrolment in the study
* At least 1 previously failed attempt to cross the CTO
* Absence of pericardial effusion on 2D Echocardiogram

Exclusion Criteria:

Candidates for this study who meet any of the following criteria at the time of the screening visit are NOT eligible to be enrolled in this study:

* Culprit vessel is a saphenous vein graft occlusion
* True ostial LAD, LCX or RCA occlusions (since collagenase delivery will be unreliable)
* Presence of moderate or large pericardial effusion on echocardiogram within 2 weeks of the procedure
* Major side branch (1.5 mm diameter) within 3 mm proximal to the occlusion. (This is to prevent the infusate being diverted through a side branch and to prevent ischemia during the prolonged period of time during the infusion)
* Renal dysfunction (creatinine greater than 2 x ULN)
* Severe calcification (collagenase can not degrade calcium) based on consensus of 2 interventional cardiologists after review of coronary angiogram.
* Subject has any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure
* Subject is a pregnant or lactating female (women of childbearing potential must have a negative serum beta-HCG within 24 hours prior to the inclusion)
* Subject is or has been partaking in another investigational product clinical study within 30 days of Screening/Day0
* Subjects with bleeding abnormalities (e.g. Factor VIII deficiency) and /or subjects that have experienced any medically documented active site of bleeding within 30 days of the screening visit, such as, but not limited to, the gastrointestinal or genitourinary tract or intercerebral hemorrhage.
* Subjects with recent acute coronary syndrome (ACS) (< 4 weeks). For those patients who had ACS ≥ 4weeks ago, only the non-culprit vessel from the recent ACS can be considered eligible for this study if all other inclusion and exclusion criteria have been met.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety | At 3 months
  * Major Adverse Cardiac events, AE and SAE.
  * Cardiac enzymes, hematology and biochemistry; changes between Screening relative to Days 1 & 30.
  * Vital Signs
  * A 2D-echocardiogram examination will be done on Day1 (18-24 hours after the collagenase administration prior to the CTO crossing procedure) and again on Day2 prior to discharge.

SECONDARY OUTCOMES:
Efficacy | Day 2
  The efficacy endpoint of this study is guidewire crossing success rates in CTOs. A response rate of 30% or greater at a particular dose will support further clinical testing of MZ-004.
Pharmacokinetic | PK blood draws will be assessed at 15, 30, 60, 120, 240, 480 min. and 18 hrs post removal of microcatheter
  Subjects in the highest dose cohort, who are participating in the PK sub-study, will have blood draws taken post dose to prior to the PCI attempt on Day2. The blood draws will coincide with standard of care blood draws, whenever possible.
  5 ml of blood will be drawn into a serum tube at each PK timepoint. All PK samples will be stored at -80 °C until the end of the study and analyzed together.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Strauss, MD, PhD, FRCP(C), Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Strauss BH, Osherov AB, Radhakrishnan S, Mancini GB, Manners A, Sparkes JD, Chisholm RJ. Collagenase Total Occlusion-1 (CTO-1) trial: a phase I, dose-escalation, safety study. Circulation. 2012 Jan 24;125(3):522-8. doi: 10.1161/CIRCULATIONAHA.111.063198. Epub 2011 Dec 16. PMID 22179536